CLINICAL TRIAL: NCT03872674
Title: A Randomized Controlled Trial Comparing High-flow Nasal Oxygen With Standard Management for Conscious Sedation During Endoscopic Retrograde Cholangiopancreatography in Prone Position
Brief Title: A Trial Comparing High-flow Nasal Oxygen With Standard Management for Conscious Sedation During Endoscopic Retrograde Cholangiopancreatography in Prone Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-2018-0082
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Patients Undergoing Endoscopic Retrograde Cholangiopancreatography in Prone Position

STUDY DESIGN:
Intervention Model Description: Arm 1: standard nasal cannula group Arm 2: high-flow humidified oxygen-delivery system (OptiFlow THRIVE) group
Masking Description: Patients will be randomly allocated to 2 groups using computer-generated randomization method. Neither participants nor physicians will be blinded to the groups because of organizational reasons
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard oxygenation(nasal cannula) (No Intervention): stand oxygenation arm will receive oxygen at 5 L/min via nasal cannula
- high-flow humidified oxygen-delivery system(OptiFlow THRIVE) (Experimental): Optiflow THRIVE arm will receive oxygen at 50 L/min via Optiflow THRIVE
  Interventions: Biological: high-flow humidified oxygen-delivery system (OptiFlow THRIVE)

INTERVENTIONS:
Biological: high-flow humidified oxygen-delivery system (OptiFlow THRIVE) — stand oxygenation arm will receive oxygen at 5 L/min via nasal cannula, while Optiflow THRIVE arm will receive oxygen at 50 L/min via Optiflow THRIVE during the procedure.
  Arms: high-flow humidified oxygen-delivery system(OptiFlow THRIVE)

SUMMARY:
Traditional conscious sedation for endoscopic retrograde cholangiopancreatography in prone position places patients at risk of desaturation, and high-flow nasal oxygen may reduce the risk. The aim of this study is to evaluate the role of high-flow nasal oxygen during endoscopic retrograde cholangiopancreatography. The investigators will compare the lowest SpO2 of standard nasal oxygen cannula group and that of high-flow humidified oxygen-delivery system group during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 1. patients who will undergo endoscopic retrograde cholangiopancreatography under conscious sedation

Exclusion Criteria:

* 1. dementia or cognitive dysfunction
* 2. altered mental status
* 3. intubated patients or tracheostomy
* 4. pregnancy
* 5. recent history of nasal bleeding
* 6. illiteracy or foreigner

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
lowest SpO2 measured with pulse oximetry during the procedure | during the procedure (from the start to the end of the endoscopic retrograde cholangiopancreatography)
  The investigators will record the lowest SpO2 during the procedure.

SECONDARY OUTCOMES:
incidence of desaturation below 90% during the procedure | during the procedure (from the start to the end of the endoscopic retrograde cholangiopancreatography)
  The investigators will compare the incidence of desaturation during the procedure between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim SH, Bang S, Lee KY, Park SW, Park JY, Lee HS, Oh H, Oh YJ. Comparison of high flow nasal oxygen and conventional nasal cannula during gastrointestinal endoscopic sedation in the prone position: a randomized trial. Can J Anaesth. 2021 Apr;68(4):460-466. doi: 10.1007/s12630-020-01883-2. Epub 2021 Jan 6. PMID 33403549